CLINICAL TRIAL: NCT04669080
Title: Developing and Evaluating an Intervention to Enhance the Work of Asthma Specialty Care Teams in Helping Families in Cost Navigation
Brief Title: Asthma Clinics Helping Expand Cost Conversations
Acronym: Asthma CHECC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Robert Wood Johnson Foundation (Other); Harvard Pilgrim Health Care (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 20-2616
Record Dates: First submitted 2020-12-07; First posted 2020-12-16 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-06

CONDITIONS: Asthma in Children
Keywords: cost of care; patient provider communication; financial burden
MeSH Terms: conditions — Financial Stress

STUDY DESIGN:
Intervention Model Description: non-randomized pre-post test
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cost navigation training intervention (Other)
  Interventions: Behavioral: Health care provider cost navigation training

INTERVENTIONS:
Behavioral: Health care provider cost navigation training — Health care providers and asthma educators in a pediatric asthma clinic will receive an online training about the importance of cost of care conversations, how to start cost of care conversations with families, how to refer families to cost navigation resources, and how to lead asthma specialty care teams in cost navigation.

SUMMARY:
Healthcare costs are a critical barrier to U.S. families' ability to access the preventive care needed to manage their children's asthma. Asthma specialty care teams are uniquely positioned to help families navigate these cost barriers, but lack structured approaches to discussing this sensitive and complex topic. This study will train asthma specialty care teams to identify families at risk for financial burden and engage in conversations about strategies to manage asthma care costs. The study team will evaluate the impact of a health care provider training on the frequency of cost navigation conversations. The investigators hypothesize that the health care provider training will increase the frequency of parent-reported cost conversations in the clinic.

ELIGIBILITY:
Inclusion Criteria:

Eligible caregivers will:

* attend a routine asthma care appointment for a 4-17 year old child
* screen positive for possible financial burden related to the cost of asthma care

Eligible healthcare providers will:

* be members of a pediatric asthma specialty care team

Exclusion Criteria:

Caregivers will not be eligible if they:

* attend an appointment for conditions other than routine asthma care
* do not screen positive for possible financial burden related to the cost of asthma care

Healthcare providers will not be eligible if they:

* are not part of the pediatric asthma specialty care team in the participating clinic

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2021-07-20 (Actual)

PRIMARY OUTCOMES:
Change in Frequency of Cost Conversations Occurring during Asthma Specialty Care Visits | Baseline, 6 weeks post intervention completion
  Change in the frequency of caregivers reporting cost of care conversations with the asthma specialty care team during routine asthma care visits

CONTACTS AND LOCATIONS:
Overall Officials: Melissa B Gilkey, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- North Carolina Children's Allergy and Asthma Center, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual quantitative data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Time Frame: 9 to 36 months following publication
Access Criteria: Investigator who proposes to use the data has IRB, IEC, or REB approval, as applicable, and an executed data use/sharing agreement with UNC.